CLINICAL TRIAL: NCT03327974
Title: Evolution of Dark Ideas When Introducing or Switching an Antidepressant: Hetero-evaluation and Use of a Smartphone Application in the Monitoring of Depression
Brief Title: Evolution of Dark Ideas When Introducing or Switching an Antidepressant
Acronym: DEPASSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem on the app, questioned the feasability of the study
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL17_0137
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Current Major Depressive Disorder
Keywords: Aged between 18 and 65; Major depressive disorder; Suicide; Ecological momentary assessment; Smartphone application
MeSH Terms: conditions — Depressive Disorder, Major; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- depressed patients (Other): All patients performed the same evaluation : ecological momentary assesement throught smartphone and 3 sheduled visits.
  All patients are depressed patients.
  Interventions: Other: DEPASSE Apllication

INTERVENTIONS:
Other: DEPASSE Apllication — Application DEPASSE in depressed patients. This application was developed by the laboratory SERVIER, by a scientific committee of psychologists and psychiatrists: Pr. Courtet, Dr Rimlinger and Pr. Swendsen.
  Depasse is available for all on the App store and on Googleplay.
  This application has several interests:
  - The first is the daily monitoring of the symptoms allowing a regular evaluation throught smileys simulating a scale from 1 to 5. The 10 parameters evaluated are: mood, dark ideas, sleep, stress, concentration, social activities, energy, pleasure, motivation and libido.
  There is the possibility to generate a graph representing the evolution of these parameters.
  Tips adapted to the actual mood are provided related to the "dysfunctional" parameters.

SUMMARY:
Depression is a frequent disease and a serious public health problem, of which suicide is the most severe complication. Its treatment is based on the introduction of antidepressant which not only proposes a significant delay in the relief of symptoms but also by the phenomenon of lifting of inhibition can increase the suicidal risk during the initiation phase. Therefore there is a major interest in proposing a monitoring of these dark and suicidal ideas, immediately after the implementation of such treatment as well as other symptoms of depression. Thus, the aim of this study is to identify the mechanisms underlying this increase in dark and suicidal ideas in this context.

DETAILED DESCRIPTION:
The study propose to assess, with an ecological momentary assessment method, the evolution of black ideas over 30 days following the introduction or switch of an oral antidepressants.

103 patients will be recruited suffering from a current major depressive disorder in the Montpellier University Hospital.

Each patient will attend a total of 3 scheduled visits, which will be completed over a period of 1 month (inclusion, between 10-15 days, 1 month. During this month, the patient will have to complete daily assesments throught a smartphone application "Depasse".

This Servier application allows the daily monitoring of symptoms allowing a regular evaluation, in the form of smileys simulating a Likert type scale evaluation of 1 to 5.

10 parameters are evaluated: moral, black thoughts, sleep, stress, concentration, social activities, energy, pleasure, motivation and libido. Note that when the patient expresses dark thoughts, he is then asked if he wants to hurt himself. If he answers yes, he is then asked to contact an emergency service.

One of its originalities is the addition of positive psychology approaches with a positive reinforcement of this evaluation through reward by a smiley in a smiley box and obtaining a "pleasant" image for motivation and incentive.

There is the possibility to have the graphical follow-up of the various parameters and to send them by mail to his treating psychiatrist.

Advice adapted to the mood of the day is provided taking into account the "dysfunctional" parameters.

Similarly, the emergency buoy tool provides access to emergency numbers and directs the patient to seek care.

Intelligence of the weight and the treatments established. The app also has a notification setting to remind the patient to evaluate themselves daily.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of a characterized depressive episode assessed by the clinician
* Depression score : MADRS> 20
* Introduction or switch of an antidepressant (without combination of molecules)
* Signed informed consent
* Able to understand the nature, purpose and methodology of the study
* French language
* Able to understand and conduct clinical assessments.

Exclusion criteria:

* The following psychiatric comorbidities: Bipolar disorder, schizophrenia, alcohol dependence and / or any other substance objectivized during the clinical evaluation
* Patient presenting a depressive episode characterized with mixed component, psychotic, melancholic or catatonic characteristics
* Score MADRS greater than or equal to 5 to one of the items
* Subject protected by law (guardianship or curatorship)
* Subject in exclusion period from another protocol
* Subject not affiliated to, or not beneficiary of, a social security scheme
* Pregnant orbreastfeeding patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Values of dark ideas assessed with a Likert type scale [1;5] | 1 month
  Evolution of dark ideas over 30 days. Throught the DEPASSE smartphone application, the patient assess the actual frequency of dark ideas from a Likert type scale of 1 (= not at all) to 5 (= often)

SECONDARY OUTCOMES:
Values of the actual mood assessed with a Lickert type scale [1;5] | 1 month
  Evolution of the mood over 30 days. Throught the DEPASSE smartphone application, the patient evaluates whether he/she is in a good mood from 1 (= not at all) to 5 (= absolutely)
Values of the actual motivation assessed with a Lickert type scale [1;5] | 1 month
  Evolution of the mood over 30 days. Throught the DEPASSE smartphone application, the patient evaluates his/her motivation from 1 (= not at all) to 5 (= absolutely)
Values of the ability to feel pleasure as usual assessed with a Lickert type scale [1;5] | 1 month
  Evolution of the mood over 30 days. Throught the DEPASSE smartphone application, the patient evaluates his/her the ability to feel pleasure as usual from 1 (= not at all) to 5 (= absolutely)
Values of the energy assessed with a Lickert type scale [1;5] | 1 month
  Evolution of the mood over 30 days. Throught the DEPASSE smartphone application, the patient evaluates whether he/she feels energetic from 1 (= not at all) to 5 (= absolutely)
Values of the social activities assessed with a Lickert type scale [1;5] | 1 month
  Evolution of the mood over 30 days. Throught the DEPASSE smartphone application, the patient assesses whether he or she is involved in social activities from 1 (= not at all) to 5 (= absolutely)
Values of the concentration assessed with a Lickert type scale [1;5] | 1 month
  Evolution of the mood over 30 days. Throught the DEPASSE smartphone application, the patient assesses his/her ability to concentrate as usual from 1 (= not at all) to 5 (= absolutely)
Values of the stress assessed with a Lickert type scale [1;5] | 1 month
  Evolution of the mood over 30 days. Throught the DEPASSE smartphone application, the patient assesses whether he feels relaxed from 1 (= not at all) to 5 (= absolutely)
Values of the libido assessed with a Lickert type scale [1;5] | 1 month
  Evolution of the mood over 30 days. Throught the DEPASSE smartphone application, if the patient has the same libido as usual from 1 (= not at all) to 5 (= absolutely)
Values of sleep assessed with a Lickert type scale [1;5] | 1 month
  Evolution of the mood over 30 days. Throught the DEPASSE smartphone application, if the patient sleep well from 1 (= not at all) to 5 (= absolutely)
Score at the Montgomery-Åsberg Depression Rating Scale (MADRS) | 1 month
  Link between the self evaluation of the patient and the evaluation conducted by the psychiatrist
Score at the Columbia Suicide Severity Rating Scale (CSSRS) | 1 month
  Link between the self evaluation of the patient and the evaluation conducted by the psychiatrist
Number of emergency room visits | 1 month
  Link between the evolution of dark ideas over 1 month and the number of emergency room visits
Number of hospitalizations | 1 month
  Link between the evolution of dark ideas over 1 month and the number hospitalizations
Satisfaction score on the Lickert type scale [1;5] | 1 month
  Assessment of the patient satisfaction regarding the utilization of DEPASSE, from 1 (= not at all) to 5 (= absolutely)

CONTACTS AND LOCATIONS:
Overall Officials: Lucile VILLAIN, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC